CLINICAL TRIAL: NCT02176044
Title: The Effect of Nitric Oxide on Spatial Working Memory in Patients With Schizophrenia - Pilot Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: NOSMEM01
Record Dates: First submitted 2014-06-25; First posted 2014-06-26 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Schizophrenia
Keywords: Nitric Oxide; Sodium Nitroprusside; Spatial Working Memory; Psychosis; Schizophrenia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucose infusion (Placebo Comparator): Placebo infusion of sterile 5% glucose - 500ml infused over 4 hours.
  Interventions: Other: Placebo
- Sodium Nitroprusside infusion (Active Comparator): Sodium nitroprusside dissolved in 5% glucose solution. Infused at 0.5mcg/kg/min for 4 hours.
  Interventions: Drug: Sodium Nitroprusside infusion

INTERVENTIONS:
Drug: Sodium Nitroprusside infusion
  Arms: Sodium Nitroprusside infusion
Other: Placebo
  Arms: Glucose infusion

SUMMARY:
Spatial working memory (ability to remember where objects are in space) is impaired in patients with schizophrenia. It is thought that this impairment occurs due to problems with the chemical messenger (neurotransmitter), glutamate, and the N-methyl-D-aspartate (NMDA) glutamate receptor, particularly in the hippocampal brain region. NMDA receptor activation leads to increases in the release of the second messenger Nitric Oxide. Impaired NMDA receptor function would therefore be predicted to lead to reductions in Nitric Oxide production. Recent work suggests that a drug, sodium nitroprusside, which releases nitric oxide, enhances some aspects of cognition in schizophrenia (specifically related to negative symptoms). In this study, the investigators will test the hypothesis that sodium nitroprusside improves spatial working memory in patients with schizophrenia. 15 patients will receive sodium nitroprusside, and 15 will receive a nonactive compound (placebo). Their performance on a spatial working memory task will be tested before and after administration of sodium nitroprusside or placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients with a diagnosis of schizophrenia or schizoaffective disorder, currently experiencing an exacerbation of symptoms (a score > 20 for PANSS-Positive subscale), currently taking antipsychotics and who have given informed consent to participate.

Exclusion Criteria:

History of hypertension or current resting systolic blood pressure greater than 140 mmHg or diastolic blood pressure greater than 90 mmHg. Relevant medical illness (renal, hepatic, cardiac), prior history of intolerance to sodium nitroprusside, presence of a seizure disorder, any change in psychotropic medication in previous 6 weeks, diagnosis of substance abuse, pregnancy (as determined by urine test) or breastfeeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Spatial Working Memory | 4 hours post-infusion
  performance on Cambridge Neuropsychological Test Automated Battery spatial working memory task

SECONDARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) | 4 hours post-infusion
  Symptoms rated on PANSS
Brief Psychiatric Rating Scale (BPRS) | 4 hours post-infusion
  Symptoms rated on BPRS
Quick Inventory of Depressive Symptomatology (QIDS) | 4 hours post-infusion
  Symptoms rated on QIDS
Hypomania Checklist (HCL-32) | 4 hours post-infusion
  Rating of symptoms on HCL-32
Blood pressure | 4 hours post-infusion
  Measurement of blood pressure.
Heart rate | 4 hours post-infusion
  Heart rate change from baseline
Respiratory rate | 4 hours post-infusion
  change in respiratory rate from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: James Stone, MBBS PhD, Principal Investigator — King's College London
Locations (1):
- Clinical Research Facility, King's College Hospital, London, United Kingdom

REFERENCES:
- [Derived] Stone JM, Morrison PD, Koychev I, Gao F, Reilly TJ, Kolanko M, Mohammadinasab A, Kapur S, McGuire PK. The effect of sodium nitroprusside on psychotic symptoms and spatial working memory in patients with schizophrenia: a randomized, double-blind, placebo-controlled trial. Psychol Med. 2016 Dec;46(16):3443-3450. doi: 10.1017/S0033291716002245. Epub 2016 Sep 22. PMID 27655012